## PROTOCOL VAN DE STUDIE

Versie 3 – 13 februari 2025

# Het Rufaida project: Onderzoek naar de impact van Ramadan vasten op het darm en vaginale microbioom

Onderzoekstudie aan de Universiteit Antwerpen, Faculteit Wetenschappen, Departement Bioingenieurswetenschappen en de Faculteit Geneeskunde en Gezondheidswetenschappen

#### Inclusie/exclusiecriteria

- Inclusiecriteria:
  - o Volwassenen van 18 jaar en ouder op het moment van inschrijving;
  - o Geslacht: vrouw;
  - o Wonend in België;
  - o Voldoende kennis van de Nederlandse taal;
  - o Toestemmingsformulier ondertekend;
- Exclusiecriteria:
  - o Menstruatie tijdens het verloop van de studie
  - o Het geven van borstvoeding bij aanvang en tijdens de studie;
  - Huidige diagnose van kanker en/of immunosuppressieve therapie in de 6 maanden voor de studie;
  - Cardiovasculaire en metabolische aandoeningen (bijvoorbeeld diabetes, prikkelbare darmsyndroom, ...);
  - o Klinisch significante neiging tot bloeden doorheen de geschiedenis;
  - o Klinisch significante afwijkingen van de voortplantingsorganen;
  - Elke andere medische aandoening die naar het oordeel van de hoofdonderzoeker aanleiding geeft tot uitsluiting van het onderzoek;
  - Gebruik van orale/vaginale antibiotica/antimycotica in de 2 maanden voor de studie:
  - o Gebruik van orale/vaginale pre-, pro- en postbiotica (i.e., supplementen bovenop de voeding) in de 2 weken voor de studie en tijdens de studie;
  - o Ketogeen dieet in de 2 weken voor de studie en tijdens de studie;
  - o Vaginaal douchen tijdens de studie;
  - o Parallelle deelname in een andere klinische studie;

## Rekrutering van participanten

De rekrutering van de vrijwilligers (minimaal n=50 voor staalafnames, n=300 voor vragenlijsten) zal verlopen via een vragenlijst die de in- en exclusiecriteria, alsook de algemene gezondheidstoestand, medicatiegebruik, etc. bevraagt. In deze vragenlijst wordt geïnformeerd of de vrijwilligers graag stalen willen afnemen of niet. Afhankelijk van hun keuze worden de

Protocol van de studie – Versie 3 – 13 februari 2025

Pagina 1 van 7

participanten in één van de twee studiepopulaties verdeeld. De vrijwilligers zullen gerekruteerd worden via verschillende kanalen, onder meer (maar niet beperkt tot) het communicatieplatform van het burgerwetenschapsproject Isala (https://isala.be/; EC nummer: B300201942076; ClinicalTrials.gov: NCT04319536) dat tot heden meer dan 6000 mensen bereikt. Indien we hiermee niet aan het vooropgestelde aantal vrijwilligers geraken, zullen andere kanalen parallel gebruikt worden voor rekrutering. Zo kunnen personeelsleden en studenten van de UAntwerpen en het UZA via affiches, ad valvas en mails uitgenodigd worden. Verder kan er ook gebruik gemaakt worden van andere kanalen, onder meer (maar opnieuw niet beperkt tot) het EOS portaal, 'Citizen Science-iedereen wetenschapper' (www.iedereenwetenschapper.be), website van de ENdEMIC (https://www.uantwerpen.be/en/research-groups/endemic/) onderzoeksgroep UAntwerpen onderzoeksgroepen, mails naar UAntwerpen geassocieerde hogescholen, andere Vlaamse universiteiten en hogescholen, nieuwe outlets, etc. Ook kan een open oproep gelanceerd worden bij deelnemers van vorige (klinische) studies uitgevoerd onder toezicht van Prof. Lebeer. Daarnaast zal er gebruik gemaakt worden van persberichten via openbare media zoals kranten en nieuwssites. Er kan ook rekrutering plaatsvinden via specifieke netwerken en organisaties, onder meer (maar niet beperkt tot) KifKif, Mahara, De Reuzen VZW, Medina Expo, etc. Verder kan de rekrutering steunen op het gekende netwerk van de betrokken arts(en), verpleegsters en dergelijke, en dit via mails, info brochures, enzovoort.

Er wordt ook een project-specifieke webpagina aangemaakt voor het Rufaida project op de Isala website (<a href="www.isala.be">www.isala.be</a>). De vrijwilligers zullen de informatie over de studie en een toestemmingsformulier ontvangen tijdens een infoavond voorafgaand aan de studie, waarbij ook de self-sampling kit verdeeld kan worden. De self-sampling kit bevat een gedetailleerde handleiding, informatiebrochure en alle materialen die de vrijwilligers nodig hebben voor de staalcollectie, -bewaring en -bezorging aan het labo van Prof. Lebeer.

# Studieverloop en staalafnames

De microbioomonderzoeken worden uitgevoerd aan de UAntwerpen, binnen het departement Bioingenieurswetenschappen in het Laboratorium van Toegepaste Microbiologie en Biotechnologie onder leiding van Prof. Dr. Ir. Sarah Lebeer. Het verloop van de studie is schematisch weergegeven in Figuur 1.



Figuur 1: Verloop van de studie.

Voorafgaand aan de studie zal een preselectiestap plaatsvinden. Deelnemers worden gevraagd om enkele vragen te beantwoorden die nagaat of ze voldoen aan de inclusie- en exclusiecriteria, waaronder een evaluatie van hun gezondheidstoestand. Indien ze worden geselecteerd, zal hun deelname aan de studie acht weken in beslag nemen. Er wordt gevraagd of ze stalen wensen af te nemen. Afhankelijk van hun antwoord worden ze in studiegroep 1 (wel stalen afnemen, n=50) of studiegroep 2 (geen stalen afnemen, n=300) geplaatst. De eerste vragenlijst zal ongeveer 35 minuten duren om in te vullen. De andere vragenlijsten zullen ongeveer 25 minuten in beslag nemen.

Voor studiegroep één (n=50) die vaginale en stoelgangstoelgang stalen zullen afnemen.

De eerste staalname vindt plaats één week voor de aanvang van de Ramadan (tijdspunt 1), waar de deelneemster ook informatie ontvangt over het gebruik van de benodigde stalen en vragenlijsten. Na het afnemen van deze stalen worden deze ingeleverd. Het tweede tijdspunt is enkele dagen voor de Ramadan (tijdspunt 2), gevolgd door een derde staalafname op tijdspunt 3. Na het afnemen van stalen van tijdspunt 2 en 3 worden deze ingeleverd. Het vierde en vijfde tijdspunt zijn gedurende de Ramadan. Na het afnemen van de stalen van tijdspunt 4 en 5 worden ze ingeleverd. De zesde staalname wordt afgenomen op het einde van de Ramadan, gevolgd door de zevende staalafname vlak na het einde van de Ramadan en de achtste staalafname een week na de Ramadan. Na het afnemen van de stalen van tijdspunt 6, 7 en 8 worden ze ingeleverd. Ieder tijdspunt wordt gepaard met een uitgebreide vragenlijst over algemene gezondheid, leefomgeving, mentale gezondheid, vaginale gezondheid, seksuele gezondheid en darm gezondheid.

Bij elk tijdspunt wordt gevraagd om (thuis) één vaginale staal en één stoelgangstoelgangstoelgang staal af te nemen, met het doeleind voor het isoleren van het DNA van de bacteriën. Na het afnemen van de stalen moeten deze direct bewaard worden in de diepvriezer (ongeveer -20°C). Daarna

moeten deze afgegeven worden in het lab van Prof. Sarah Lebeer (Campus Groenenborger, gebouw V, verdieping 5, adres: Groenenborgerlaan 171, 2020 Antwerpen).

Bij tijdspunt 1, 3, 5 en 8 wordt gevraagd om (thuis) één additionele vaginale en één additionele stoelgangstoelgangstoelgang staal af te nemen, deze worden gebruikt om te achterhalen welke extra producten dat de micro-organismen maken aanwezig zijn in het milieu. Na het afnemen van de stalen moeten deze direct bewaard worden in de diepvriezer (+/- -20°C). Daarna moeten deze afgegeven worden in het lab van Prof. Sarah Lebeer (Campus Groenenborger, gebouw V, verdieping 5, adres: Groenenborgerlaan 171, 2020 Antwerpen).

Voor studiegroep twee (n=300) die enkel vragenlijsten zullen invullen.

Op elk tijdspunt zal de deelneemster een mail krijgen met een vragenlijst over algemene gezondheid, leefomgeving, mentale gezondheid, vaginale gezondheid, seksuele gezondheid en darm gezondheid

De verwerking en analyse van de stalen zal plaatsvinden onder leiding van de UAntwerpen, binnen het departement Bio-ingenieurswetenschappen in het labo van Prof. Sarah Lebeer. We zullen het genetisch materiaal van de micro-organismen uit de stoelgangstoelgang en vaginale stalen isoleren en kijken naar welke producten geproduceerd worden. Dit helpt ons om de algemene gezondheid te begrijpen en hoe de darm- en vaginale microbiomen met elkaar samenwerken.

stoelgangstoelgang

Door deze gestructureerde aanpak hopen we inzicht te krijgen in de impact van Ramadan vasten op de micro-organismen die aanwezig zijn in de darmen en de vagina, en welke gevolgen dit kan hebben daarvan voor de gezondheid van vrouwen. Na het aflopen van de studie zal de participant van ons een analyse krijgen van hun persoonlijk microbioom met een woordje uitleg over de bacteriën die we hebben gevonden. Op een later tijdstip zal er ook een algemene communicatie zijn over de resultaten van de studie.

#### Steekproefgrootte berekening

Power-analyses vormen een grote uitdaging voor microbioomstudies. Dit komt doordat de grootte en variantie van de effecten onbekend zijn, daarenboven ook sterk afhankelijk van het individu en bovendien voor bacterie verschillend. Om de hoeveelheid deelnemers te bepalen baseren we ons op gelijkaardige studies die het effect van intermittent fasting zoals de Ramadan op het microbioom onderzoeken. Bijvoorbeeld, in de cross-sectional study door Mohammed-zadeh *et al.* (2021) werden stoelgangstalen van 30 participanten verzameld voor en na de Ramadan, om het effect van vasten op het darm microbioom te onderzoeken. Dit was voldoende om veranderingen in het microbioom waar te nemen tijdens het vasten verlaagt. Studies die het darm microbioom tijdens de Ramadan analyseerde hadden van 9 (Ozkul *et al.* 2020) tot 67 deelnemers (Ali *et al.* 2021). Naar ons beste weten zijn er nog geen studies uitgevoerd die het effect van Ramadan vasten op het vaginale en darm microbioom onderzochten. Daarom kiezen wij om 50 vrijwilligers te includeren om de vragenlijsten in te vullen en de stalen af te nemen, en 300 vrijwilligers om de vragenlijsten

Gewijzigde veldcode

Gewijzigde veldcode

in te vullen zonder stalen af te nemen. In de voorgaande fase van het Rufaida project (enkele vragenlijsten) waren 245 participanten geregistreerd.

### Analyse van de stalen

Labo Toegepaste Microbiologie en Biotechnologie Prof. Sarah Lebeer, Faculteit Wetenschappen, Departement Bio-ingenieurswetenschappen, UAntwerpen

#### Deel 1: Microbioomanalyse

Microbieel DNA zal geïsoleerd worden van verschillende lichaamslocaties en -vloeistoffen (vaginale wisser, fecaal staal en urine container). De samenstelling van de microbiële gemeenschap (bacteriën, virussen, schimmels, etc.) zal worden geanalyseerd op basis van het genetisch materiaal van deze microbiële gemeenschap aanwezig in de verzamelde stalen. Hiervoor zal het totale DNA van de stalen geïsoleerd worden via commercieel beschikbare DNA-extractie-kits (bv. Qiagen PowerFecal PRO of Qiagen PowerSoil PRO DNA kit of gelijkaardig). Het geïsoleerde DNA zal vervolgens geanalyseerd worden via amplicon en shotgun sequenering (bv. Illumina en Nanopore sequencing platforms) om zo specifiek mogelijk de aanwezige micro-organismen en hun genomen in kaart te brengen. Het geïsoleerde DNA zal vervolgens geanalyseerd worden via amplicon sequenering (gebaseerd op het 16S rRNA gen) en shotgun sequenering. Het 16S rRNA gen bestaat uit 9 verschillende variabele regio's, die gebruikt kunnen worden voor de microbiële karakterisatie en die geflankeerd worden door geconserveerde regio's. Deze laatste worden als target gebruikt voor 'polymerase chain reaction' (PCR)-primers met een universele specificiteit voor bijna alle bacteriën. Er zal gebruik gemaakt worden van het Illumina sequencing platform bij een externe partner (bijvoorbeeld Prebiomics) en in het Centrum voor Medische Genetica. Het protocol voor microbioomanalyse van humane stalen werd geoptimaliseerd in de onderzoeksgroep (Ahannach et al., 2021) en zal in deze studie geïmplementeerd worden.

**Mijlpaal:** Identificatie van verschillen in de microbioomsamenstelling van de verschillende lichaamslocaties en -vloeistoffen van de vrijwilligers

## Deel 2: Kwantitatieve analyse van concentratie specifieke micro-organismen

Via "quantitative real-time polymerase chain reaction" (qPCR) zal m.b.v. stam-, species- of genus-specifieke primers de concentratie van bepaalde micro-organismen. Bij qPCR wordt de hoeveelheid van een specifiek stuk DNA in 'real time' gemeten. Hierdoor kan de initiële concentratie van dit specifiek DNA bepaald worden. De resultaten geven zo dan een beeld over de concentratie van verschillende micro-organismen in een staal. Voor de verwerking van deze data zullen de "Minimum Information for Publication of Quantitative Real-Time PCR Experiments" (MIQE) richtlijnen gebruikt worden, zoals beschreven (Bustin et al., 2009).

**Mijlpaal:** Absolute abundantie van micro-organismen in verschillende lichaamslocaties en -vloeistoffen van de vrijwilligers

Deel 3: Cultiveren van melkzuurbacteriën en andere beneficiaire micro-organismen uit vaginale stalen

De huidige probiotische stammen, meestal melkzuurbacteriën, zijn typisch geïsoleerd van de gastro-intestinale niche van ons lichaam. Voor toepassingen van probiotica in de vagina zou het echter interessant zijn om melkzuurbacteriën te isoleren uit de vagina. Hierbij is het verwacht voordeel dat niche-specifieke stammen beter zijn aangepast aan de condities in de vagina en beter zijn opgewassen tegen de daar ook aanwezige pathogene bacteriën. Melkzuurbacteriën zijn interessant omdat ze een GRAS status hebben ('Generally Recognized As Safe') en talrijke gezondheidseffecten uitgebreid zijn beschreven, maar ook omdat recente studies hebben aangetoond dat lagere hoeveelheden melkzuurbacteriën gepaard gaan met meer vaginale infecties. Bijgevolg zullen we vaginale wissers van de vrijwilligers uitplaten op selectieve media voor melkzuurbacteriën, zoals MRS (de Man Rogosa and Sharpe), LAMVAB medium en bloedagar. Hiervoor zal de wisser opgelost worden in PBS (Phosphate Buffered Saline) en na grondig mengen zal een verdunningsreeks uitgeplaat worden. Verschillende kolonies zullen aangestipt worden en verdere identificatie op species level zal gebeuren via kolonie-PCR met universele primers voor het *16S rRNA* gen (bijvoorbeeld 8F-1525R), gevolgd door Sanger sequenering en alignatie t.o.v. een referentiegenoom (bijvoorbeeld d.m.v. BLAST, EZBioCloud of een in-house pipeline).

Mijlpaal: Cultiveren van minimum 50 vaginale melkzuurbacteriën

#### Deel 4: Identificatie en kwantificatie van metabolieten uit wissers/lichaamsvloeistoffen

Naast de identificatie en kwantificatie van specifieke micro-organismen uit wissers en staalnames is het ook interessant om te kijken naar welke metabolieten geproduceerd worden door deze micro-organismen en in welke concentratie. Dit kan achterhaald worden met behulp van metabolomics. Concreet zal ("Ultra-high performance") vloeistofchromatografie en (hoge-resolutie) massaspectrometrie toegepast worden op de afgenomen stalen/supernatans van oplossingen die verder zullen bereid worden door extractie met een koud organisch oplosmiddel na toevoeging van een intern standaardmengsel. Geschikte software (bijvoorbeeld de MassHunter Quantitative/Qualitative Analysis Software) zal vervolgens worden gebruikt voor identificatie en kwantificatie van metabolieten, gevolgd door piekuitlijning, waardoor metabolietannotatie en statistische analyses mogelijk zijn. Vervolgens zal de data aan de hand van bio-informatische hulpmiddelen verder geanalyseerd en gevisualiseerd worden. Naast deze microbieel geproduceerde metabolieten zullen ook metabolieten afkomstig van de voeding, de omgeving en dergelijke bestudeerd worden met bijbehorende identificatie en/of kwantificatie.

Wat betreft de korte-keten vetzuren zal de modulatie van lokale levels onderzocht worden in vaginale wissers en stoelgangstoelgangstoelgang stalen. Dit zal gebeuren aan de hand van (un)targeted metabolomics analyse met technieken zoals massaspectrometrie (LC-MS en GC-MS) om zo het verdere effect op het microbioom, metaboloom en de algemene gezondheid te bepalen.

**Mijlpaal:** Identificatie en kwantificatie van metabolieten in verschillende lichaamslocaties en vloeistoffen van de vrijwilligers, met een gerichtere focus op riboflavine en korte-keten vetzuren

## Referenties

Ahannach, S., Delanghe, L., Spacova, I., Wittouck, S., Van Beeck, W., De Boeck, I., & Lebeer, S. (2021). Microbial enrichment and storage for metagenomics of vaginal, skin, and saliva samples. *iScience*, 24(11), 103306. https://doi.org/10.1016/j.isci.2021.103306

Bustin, S. A., Benes, V., Garson, J. A., Hellemans, J., Huggett, J., Kubista, M., Mueller, R., Nolan, T., Pfaffl, M. W., Shipley, G. L., Vandesompele, J., & Wittwer, C. T. (2009). The MIQE guidelines: minimum information for publication of quantitative real-time PCR experiments. *Clinical chemistry*, 55(4), 611–622. https://doi.org/10.1373/clinchem.2008.112797

Ozkul, C., Yalinay, M., & Karakan, T. (2020). Structural changes in gut microbiome after Ramadan fasting: A pilot study. *Beneficial Microbes*, 11(3), 227–233. https://doi.org/10.3920/BM2019.0039

Mohammadzadeh, A., Roshanravan, N., Mesri Alamdari, N., Safaiyan, A., Mosharkesh, E., Hadi, A., Asghari Jafarabadi, M., & Meshkani, R. (2021). The interplay between fasting, gut microbiota, and lipid profile. *International Journal of Clinical Practice*, 75(10), e14591. https://doi.org/10.1111/jjcp.14591

Ali, I., Madkhali, N., Alreshidi, M., & Siddiqui, M. A. (2021). Ramadan fasting leads to shifts in human gut microbiota structured by dietary composition. *Frontiers in Microbiology*, *12*, 642999. https://doi.org/10.3389/fmicb.2021.642999